CLINICAL TRIAL: NCT01662609
Title: Protocol for High-Risk Assessment, Screening, and Early Detection of Pancreatic Cancer at Moffitt Cancer Center and Lehigh Valley Hospital
Brief Title: Protocol for High-Risk Assessment, Screening, and Early Detection of Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-14882
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer
Keywords: pancreas; high-risk
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endoscopic Ultrasound (EUS) Participants: High-risk for Pancreatic Cancer: Patients with 2 or more relatives with pancreatic cancer and a first degree relationship with at least one of the relatives with pancreatic cancer.
  Interventions: Procedure: Endoscopic Ultrasound (EUS)

INTERVENTIONS:
Procedure: Endoscopic Ultrasound (EUS) — Ultrasound scope will be passed through the participant's mouth into their stomach and their pancreas will be evaluated completely by the ultrasound scope. If an abnormality is found in their pancreas, a biopsy may be performed to obtain a diagnosis.
  Other Names: ultrasound scope

SUMMARY:
The purpose of this study is to find out whether Endoscopic Ultrasound (EUS) can detect early stage pre-cancerous or cancerous changes in the pancreas in patients at high-risk for the development of pancreatic cancer. Endoscopic refers to the use of an instrument called an endoscope - a thin, flexible tube with a tiny video camera and light on the end. Ultrasound refers to an imaging technique that uses sound waves to produce pictures. EUS in this research study is a method of combining endoscopy and ultrasound imaging to obtain high quality images of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they have 2 or more relatives with pancreatic cancer and have a first degree relationship with at least one of the relatives with pancreatic cancer

  * If only 2 family members are affected then both must have had pancreatic cancer and a first-degree relationship with individual screened
  * If there are more than 2 affected individuals on the same side of the family at least one of the individuals must have a first-degree relationship with the member being screened
  * Patients at least 40 years old or 10 years younger than the youngest affected individual
* Peutz-Jeghers Syndrome (PJS) patients age>30
* Hereditary pancreatitis patients
* Patients with Familial Atypical Multiple Mole Melanoma Syndrome (FAMMM)
* Patients with BRCA2 mutation and at least one first or second degree relative with documented pancreatic cancer
* Willingness to undergo (EUS) with possible Fine Needle Aspiration (FNA)
* Willingness to undergo surgical evaluation for abnormal EUS/FNA finding
* Willingness to undergo radiographic evaluation if screening findings are abnormal

Exclusion Criteria:

* Medical contraindications to undergoing endoscopy or obstruction of the GI tract that precludes passage of the endoscope
* Personal history of pancreatic adenocarcinoma
* Previous partial or complete resection of the pancreas for adenocarcinoma
* Prior partial or total gastrectomy with Billroth II or Roux-en-Y anastamosis
* Previous computed tomography (CT) scan, magnetic resonance imaging/magnetic resonance cholangiopancreatography (MRI/MRCP) or EUS of the abdomen in the past 3 years
* Coexisting cancer in other organs or acquired immunodeficiency syndrome/human immunodeficiency virus (AIDS/HIV)
* Life expectancy less than 5 years
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals potentially at high-risk for developing pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2007-08-23 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Number of Abnormalities Detected by EUS | Average of 5 years
  To determine whether targeted screening of these high-risk individuals using Endoscopic Ultrasound (EUS) at regular intervals can detect precancerous pancreas changes or early stage asymptomatic pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Dam, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/